CLINICAL TRIAL: NCT06740279
Title: Investigating the Upper Limb During the First 6 Months After Sustaining a Cervical Spinal Cord Injury,
Acronym: In Ul 6 SCI
Status: Not yet recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Promobilia Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: InUL6SCI; ALFGBG-984319 (Other: VästraGötalandsregionen); 282763 (Other: https://www.researchweb.org/is/sverige/project/282763)
Record Dates: First submitted 2024-12-09; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries (SCI); Upper Limb Function
Keywords: Spinal cord injury; Upper limb; tetraplegia; Quadriplegia; hand function; Activities of daily living; grip ability
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment of upper limb function — Observational study of the changes in upper limb after SCI paralysis

SUMMARY:
The goal of this observational study is to investigate and describe the injury patterns, secondary complications, and biomechanical properties of the upper limb during the initial 6 months post-SCI.

The overarching objective is to investigate and describe the trajectory of upper limb functioning, secondary complications, and biomechanical properties of the upper limb during the initial 6 months post-SCI and explore factors influencing functional use of the hands at 6 months after injury.

DETAILED DESCRIPTION:
INTRODUCTION Sustaining a cervical spinal cord injury (SCI) leads to tetraplegia with paralysis in all four extremities. It is a traumatic event that radically changes an individual's ability to perform activities of daily life. Our arms and hands are critical functions since most of our daily activities depend on our hands. A person with tetraplegia also needs the upper limb (UL) to compensate for the paralysed legs in activities such as wheelchair mobility and transfers. Recovery of hand function has in several studies been depicted as the most important function to recover by people with tetraplegia.

Despite the importance of hand function, the evidence for treatment and optimization of the UL after tetraplegia is underdeveloped. Intervention studies targeting the tetraplegic UL typically focus on a single intervention and individuals in a chronic stable phase. The international clinical experience is that there are known factors that has the potential to impact the UL after c-SCI and studies investigating the incidence, timeframes and potential consequences for a functional UL in the acute and early phase are lacking.

Aim/Study rationale The overarching objective is to develop and assess a structured treatment plan for upper limb rehabilitation following cervical spinal cord injury (SCI). The ultimate aim is to empower patients with functional hands that enable daily living activities, emphasizing optimized grip strength and minimal range of motion limitations.

To achieve this, it is crucial to thoroughly investigate and describe the injury patterns, secondary complications, and biomechanical properties of the upper limb during the initial 6 months post-SCI.

METHODS Data collection and study sites This is a prospective cohort study. The study is designed to cover the absolute majority of people sustaining a cervical SCI during one year in Sweden and New Zealand. Inclusion criteria is to be found in the study design section. Following study sites will be included; in Sweden; Region Skåne, Region Västerbotten, Region Stockholm, Västra Götalandsregionen. In New Zealand, the two national spinal units in Auckland and Christchurch. Additional data will be collected from Lyndhurst Toronto rehab, KITE, Toronto, Canada. The Swiss Paraplegic Center, Notwill Switzerland will also be involved. Data will be collected at 1,2,3 and 6 months after sustained c-SCI. When available, additional assessment 1-2 weeks after injury will be included. The study aims to recruit patients for one year.

Sample size The sample size is not based on a formal sample size calculation, since this is an exploratory study investigating the injury pattern and its consequences related to the upper limb. With several assumptions due to lack of comprehensive data the estimated total number is 210 participants (420 arms) to be included and 140 participants (280 arms) to be included in the 6 months follow up. Approximately 420 arms is considered to be a feasible number to secure the primary research question; describe the injury pattern. For the secondary question, were the 6 months follow up is crucial a total of 280 arms is considered sufficient to adequately test for interactions.

Datacollection Assessment will be done by training Occupational therapists at 1 ,2, 3 (+-1w) months and 6 months (-1+2months). A detailed description of the data collection in an examiners manual will be available and all site investigators will receive specific training prior study start to secure required competence and measuring alinements between the sites. The Coordinating investigator (PI) will commence regular meetings (approximately once a month) and also chat function together with the site investigators to secure forums to clarify any questions during the data collecting phase. Outcome measures and timepoints for each measure in the study is to be found in the outcome measure section.

Site investigator verifies that each patient has consented to direct access to the original source data/hospital records, by the use of written patient information and signed Informed consent. Thereafter the site investigator will register coded original source data into the electronic system RedCap that is provided by the Coordinating investigator through Västra Götalands regionen, who is also responsible for the system. All information processed by the PI and steering group will be pseudonymized and identified with a study code. Subjects will not be identified by their names, but by an identification code in RedCap, and in other relevant study documents.

Data analysis Sahlgrenska University Hospital (SUH), as part of Region Västra Götaland, is the entity responsible for research and Personal Data Controller and will store the RedCap system (the eCRF-system used in the study). SUH will also be in charge of the statistical analyses and will be a Personal Data Processor in the study.

Demographics and timepoint specific characteristics will be summarized descriptively and changes over time will be described. Descriptive statistics that will be presented are number of observations and proportions for categorical variables, and number of observations, means, standard deviations, medians, quartiles and ranges for continuous variables.

Linear regression will be used to investigate whether the functional outcome (GRASSP, SCIM and TUAQ) is dependent on baseline characteristics. The Jonckheere-Terpstra test will be used to determine if there is a statistically significant trend between ordinal independent variables and a continuous or ordinal dependent variables. All tests will be two-tailed and conducted at 0.05 significance level.

The exact co-variates will be defined in the statistical analysis plan (SAP) and will include e.g.:

* Age
* Sex
* Severity of injury (ISNCSCI; C1,C2, C3, C4, C5, C6, C7) (AIS; A,B,C,D)
* Secondary complications (stiffness; prevalence of restrictions over 20 degrees,) (spasticity; prevalence of MAS 0, 1-2 and 3-4) (swelling; prevalence of increased circumference >1cm )
* Remaining motor function (total number of innervated muscles (1-5), total number of muscles >MRC 3, grouping data into flexors and extensors)
* Motor excitability (number of innervated muscles (=2), partly denervated muscles (=1) and denervated muscles (=0), grouping data into flexors and extensors.
* Biomechanical properties (resting position, hand opening/closing and pinch opening/closing, respectively; 0= no/minimal opening/closing, 1= some but not functional, 2= over half opening/closing, 3=3/4 open/closing, 4=normal) Multivariate analyze will be used to investigate explanatory factors to grip ability (GRASSP) and patients' satisfaction with grip ability (TUAQ) at 6 months. The aim is to assess differences between sub-groups with respect to the secondary endpoints using Cox regression models including Grip ability variable and subgroup factor and also the interaction between these variables as independent variables will be tested. The subgroups will be based on for example sex, age, injury severity, secondary complications, biomechanical properties and will be further pre-specified in the SAP.

Categorical endpoints will be analyzed using unadjusted and adjusted logistic regression models. Odds ratios (OR) and 95% CIs will be presented. Linear models will be used to analyze continuous variables, with logarithmic transformations applied if needed. Mean values and 95% CIs and OR will be presented.

Prior to start of data analysis, a separate statistical analysis plan (SAP) describing the intended statistical analyses and derivation of variables in greater detail, will be finalized.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Acute onset Cervical SCI (traumatic and non-traumatic) C0-C7 AIS A-D that affects motor function in the upper limb.
* Over the age of 18 at admission
* Admitted for rehabilitation at one of the study sites.

Exclusion Criteria:

* For the surveys: Inability to understand Swedish or English in writing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals with acute onset cervical SCI (traumatic and non-traumatic) C0-C7 AIS A-D that affects motor function in the upper limb at the following study sites will be invited; In Sweden; Region Skåne, Region Västerbotten, Region Stockholm, Västra Götalandsregionen.
  In New Zealand, the two national spinal units in Auckland and Christchurch. In Canada: Lyndhurst Toronto rehab, KITE, Toronto.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2025-01-07 (Estimated); Primary Completion 2026-10-06 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Motor neuron testing | 1,2,3,6 months post injury
  Motor neuron testing, using the well established NeuroMuscular Electrical Stimulation (NMES). Identification of the LMN integrity in defined muscle will be done by surface electrical stimulation of the forearm according to standardized technique (Bersch 2018). A standard four-channel nerve stimulator ( Chattanooga Rehab SKU 2533110-INT) will be used and with stimulation parameters according to international recommendations for nerve/muscle stimulation; 20-80 mA, 250-300 μs at 35 Hz (Bersch 2022). All stimulators have CE approval, approved as medical technical product (medicinteknisk produkt) in Sweden and manuals in both Swedish and English are available. The stimulator will be used within approved area.

OTHER OUTCOMES:
International Standards for Neurological Classification of SCI (ISNCSCI) including the American Spinal Injury Association Impairment Scale (AIS) | At admission and discharge from inpatient setting. Both assessments will be from date of inclusion until the date of final assessment at 6 months (-1+2 months) or date withdrawn from study, whichever came first, assessed up to 8 months
  ISNCSCI and AIS are well-established international communication tools for researchers and clinicians to quantify the neurological impairment resulting from a spinal cord injury. (Kirshblum 2011) The ISNCSCI examine the motor- and sensory level of injury, C1- C7. While the AIS describe the completeness of the injury using a 5-point ordinal scale, classifying individuals from A" (complete SCI) to "E" (normal sensory and motor function) The ISNCSCI and AIS is part of clinical routine at admission and discharge
Muscle strength | 1,2,3,6months
  Active motor strength, as measured by the Medical Research Council are considered golden standard for muscle testing.
Modified Ashworth scale | 1,2,3,6 months
  Modified Ashworth scale (Baunsgaard 2016) is considered one of the golden standard measures in measuring spasticity in SCI. The scale go from 0-5 where 0=no spasticity and 5=rigid.
Biomechanical balance of the hand | 1,2,3,6 months
  Observation of the maximal hand opening and closing.
Swelling of the hand | 1,2,3,6 months
  Swelling will be assessed with a measuring tape according to the figure of eight, which is a valid and reliable assessment of swelling in a hand (Shaban 2013)
Spinal Cord Independence Measure, SCIM-SR | admission, discharge, Both assessments will be from date of inclusion until the date of final assessment at 6 months (-1+2 months) or date withdrawn from study, whichever came first, assessed up to 8 months. And 6 months
  The SCIM is the internationally the most common measure for level of independence after SCI. The newly validated Swedish version (Jörgensen 2021) is a part of an ongoing study in most sites in Sweden at 1 and 12 months and part of clinical routine in Switzerland and New Zealand at admission and discharge. This study will use the self report, SCIM-SR.
Tetraplegia Upper limb Activity Questionnaire, TUAQ: | admission, discharge,Both assessments will be from date of inclusion until the date of final assessment at 6 months (-1+2 months) or date withdrawn from study, whichever came first, assessed up to 8 months. And 6 months
  The TUAQ is a questionnaire specific for skilled hand use for the tetraplegic population and gives the patients perspective of their ability to use their hands in daily life (Wangdell 2022 x2) . The TUAQ is validated in Swedish and English (Wangdell 2022).
Graded Redefined Assessment of Strength, Sensibility, and Prehension, GRASSP part 2. | 1,2,3,6months
  The GRASSP is the internationally most commonly used hand assessment in acute SCI. Part 2 quantifies patients' ability to grasp and use the hand in activities by assessing the ability to handle 6 different objects (Kalsi-Ryan 2012).

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Wangdell, PhD, Principal Investigator — Västra Götalandsregionen, Sahlgrenska University Hospital

IPD SHARING:
Plan to Share IPD: No
Data will only be analysed on group level and within the research group.

REFERENCES:
- [Result] Harvey LA, Dunlop SA, Churilov L, Hsueh YS, Galea MP. Early intensive hand rehabilitation after spinal cord injury ("Hands On"): a protocol for a randomised controlled trial. Trials. 2011 Jan 17;12:14. doi: 10.1186/1745-6215-12-14. PMID 21235821
- [Result] Anderson KD. Targeting recovery: priorities of the spinal cord-injured population. J Neurotrauma. 2004 Oct;21(10):1371-83. doi: 10.1089/neu.2004.21.1371. PMID 15672628
- [Result] Grampurohit N, Bell A, Duff SV, Mulcahey MJ, Thielen CC, Kaplan G, Marino RJ. Highlighting gaps in spinal cord injury research in activity-based interventions for the upper extremity: A scoping review. NeuroRehabilitation. 2021;49(1):23-38. doi: 10.3233/NRE-210042. PMID 33967071
- [Result] Snoek GJ, IJzerman MJ, Hermens HJ, Maxwell D, Biering-Sorensen F. Survey of the needs of patients with spinal cord injury: impact and priority for improvement in hand function in tetraplegics. Spinal Cord. 2004 Sep;42(9):526-32. doi: 10.1038/sj.sc.3101638. PMID 15224087
- [Result] Baunsgaard CB, Nissen UV, Christensen KB, Biering-Sorensen F. Modified Ashworth scale and spasm frequency score in spinal cord injury: reliability and correlation. Spinal Cord. 2016 Sep;54(9):702-8. doi: 10.1038/sc.2015.230. Epub 2016 Feb 9. PMID 26857270
- [Result] Kirshblum SC, Burns SP, Biering-Sorensen F, Donovan W, Graves DE, Jha A, Johansen M, Jones L, Krassioukov A, Mulcahey MJ, Schmidt-Read M, Waring W. International standards for neurological classification of spinal cord injury (revised 2011). J Spinal Cord Med. 2011 Nov;34(6):535-46. doi: 10.1179/204577211X13207446293695. No abstract available. PMID 22330108
- [Result] Bersch I, Koch-Borner S, Friden J. Electrical stimulation-a mapping system for hand dysfunction in tetraplegia. Spinal Cord. 2018 May;56(5):516-522. doi: 10.1038/s41393-017-0042-2. Epub 2018 Jan 22. PMID 29358674
- [Result] Bersch I, Krebs J, Friden J. A Prediction Model for Various Treatment Pathways of Upper Extremity in Tetraplegia. Front Rehabil Sci. 2022 Jun 30;3:889577. doi: 10.3389/fresc.2022.889577. eCollection 2022. PMID 36188973
- See also: Swedish research database. English title:Investigating the upper limb during the first 6 months after sustaining a cervical spinal cord injury — https://www.researchweb.org/is/sverige/project/282763